CLINICAL TRIAL: NCT04658888
Title: Increasing Cervical Cancer Screening Among Female Patients at Penn State Health St. Joe's Residency Clinic: Letter Notifying Them About Outdated Screen and Postcard With Self-sampling Option
Brief Title: St. Joe's Invitation Effectiveness Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Christina Scartozzi, Assistant Professor, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 14823
Record Dates: First submitted 2020-11-30; First posted 2020-12-09 (Actual); Results first posted 2022-07-06 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-06

CONDITIONS: Cervical Cancer Screening
Keywords: Cervical Cancer; Self-Sampling
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Intervention Model Description: This study will use a two armed model: an intervention and a control arm. The control arm will use a standard of care letter reminding the participant to schedule their screening with their primary care provider. The intervention arm will consist of a modified letter with a postcard giving the participant the option to request a self-sampling kit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Modified letter with self-sampling request card (Experimental): This group will receive a modified letter telling the participant they are out of date with their cervical cancer screening. They will also receive information on the self-sampling kit and will be provided a card that they can send back to the study team in order to have a kit sent to their house. The kit will include a pre-paid mailer so that it can be sent back to the lab for testing. The result will then be shared with the participant.
  Interventions: Device: Evalyn Self-Sampling Brush
- Standard letter (No Intervention): Participants will receive a standard of care letter that tells the participant they are out of date with their cervical cancer screening and should contact their primary care provider to schedule an appointment.

INTERVENTIONS:
Device: Evalyn Self-Sampling Brush — A self-sampling brush to collect cervical cancer cells for screening purposes.
  Arms: Modified letter with self-sampling request card

SUMMARY:
The objective of this study is to evaluate the effectiveness of offering self-sampling for high risk human papilloma virus (HPV) testing in order to increase the number of women who are screened for cervical cancer. The hypothesis of this study is that women who are notified of a need for cervical cancer screening by letter and are also offered a self-sampling kit for cervical cancer screening will have a higher rate of screening than women notified by letter alone.

This study will use an intervention arm (letter and option to request a self-sampling kit) compared to a control arm (letter alone, standard of care) as a reminder that they are out of date for their cervical cancer screening. Women who are out of date with their cervical cancer screening will be identified using the Electronic Medical Record and randomized to the study group in a 2 to 1 ratio (2 for the control arm and 1 to the intervention arm). The primary endpoint that will be evaluated in this study is the method of completion of cervical cancer screening and the use of the self-sampling kit, which will be monitored over a three month period after the letters have been mailed. A secondary endpoint will be the overall rate of cervical cancer screening of all people mailed a letter.

DETAILED DESCRIPTION:
The American Cancer Society estimates that 4,170 women in the United States will die from cervical cancer in 2018. It is possible to prevent many of these deaths through screening and appropriate follow-up in women with positive screens (1). Self-sampling for HPV testing may be a viable option for cervical cancer screening, particularly among women who do not obtain regular screening in a clinical setting.

The objective of this study is to evaluate the effectiveness of offering self-sampling for high risk HPV testing to in order to increase the number of women who are screened for cervical cancer at the Penn State Health (PSH) St. Joseph's family and community medicine residency clinic. This study will use an intervention arm and a control arm. Women in the control arm will receive a standard letter stating that they need to be screened and should contact their primary care provider. Women in the intervention arm will receive a modified version of the letter informing them of a self-sampling option with a pre-addressed post card that allows them to request a self-sampling kit. Once the postcard is returned these women will receive a self-sampling kit in the mail to collect their sample. The kit will come with a pre-paid mailer so that the participant can return their kit for processing at the Penn State Hershey Clinical laboratory.

Women who are out of date with their cervical cancer screening will be identified using the Electronic Medical Record by the use of a set of queries that have been developed to extract this patient population. Eligible women will be randomized to the study group in a 2 to 1 ratio (2 for the control arm and 1 to the intervention arm). The primary endpoint that will be evaluated in this study is the method of completion of cervical cancer screening and the use of the self-sampling kit, which will be monitored over a three month period after the letters have been mailed. A secondary endpoint will be the overall rate of cervical cancer screening of all people mailed a letter. Participants will be recruited continuously until the anticipated sample size has been met. A total of 1,211 participants are expected to participate in this study, 807 in the control arm and 404 in the intervention arm. The study team will calculate the proportion of participants who obtain cervical cancer screening from the clinic or the self-sampling kit and use chi-square tests for statistical analysis.

If a self-collected cervical sample produces a negative result, the participant will be contacted by a study physician with these results. If the sample produces a positive result for low-risk HPV the participant will be contacted by a study physician to schedule a pap test. If the sample produces a positive result for high-risk HPV the participant will be contacted by a study physician for a colposcopy. The pap test and colposcopy are both standard of care for these results. The study team will monitor the completion of the screenings and subsequent procedures.

ELIGIBILITY:
Inclusion Criteria:

* Female patients at Penn State Health St. Joe's Family and Community Medicine residency clinic or women's health clinic.
* Ages 30-65 years
* Out-of-date for cervical cancer screening
* Able to speak, read, and communicate well in English or Spanish
* Not greater than average risk for cervical cancer screening

Exclusion Criteria:

* Pregnant
* Incarcerated
* Greater than average risk for cervical cancer (2)
* Have a compromised immune system
* With in-utero exposure to diethylstilbestrol
* Unable to speak, read, and communicate well in English or Spanish
* Unable or unwilling to give implied consent or otherwise complete study requirements

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 964 (Actual)
Dates: Start 2021-04-26 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christina Scartozzi, DO, Principal Investigator — Penn State College of Medicine
Locations (1):
- Penn State College of Medicine, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2018. CA Cancer J Clin. 2018 Jan;68(1):7-30. doi: 10.3322/caac.21442. Epub 2018 Jan 4. PMID 29313949
- [Background] US Preventive Services Task Force; Curry SJ, Krist AH, Owens DK, Barry MJ, Caughey AB, Davidson KW, Doubeni CA, Epling JW Jr, Kemper AR, Kubik M, Landefeld CS, Mangione CM, Phipps MG, Silverstein M, Simon MA, Tseng CW, Wong JB. Screening for Cervical Cancer: US Preventive Services Task Force Recommendation Statement. JAMA. 2018 Aug 21;320(7):674-686. doi: 10.1001/jama.2018.10897. PMID 30140884

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A report from the electronic medical record identified woman ages 30-65 who were out of date for cervical cancer screening. Letters were sent to the patient's home during June-July 2021.
Pre-assignment Details: No participants who qualified were excluded from the study.
Groups:
- Modified Letter With Self-sampling Request Card: This group received a modified letter telling the participant they are out of date with their cervical cancer screening, received information on the self-sampling kit and postcard to request a kit.
- Standard Letter: Participants received a standard of care reminder letter telling the participant they are out of date with their cervical cancer screening and to contact their primary care provider to schedule an appointment.
Period: Overall Study
Arm/Group | Modified Letter With Self-sampling Request Card | Standard Letter
Started | 333 | 631
Completed | 333 | 631
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Modified Letter With Self-sampling Request Card: This group received a modified letter telling the participant they are out of date with their cervical cancer screening. They also received information on the self-sampling kit and were provided a card that they can send back to the study team in order to have a kit sent to their house. The kit included a pre-paid mailer so that it can be sent back to the lab for testing.
  Evalyn Self-Sampling Brush: A self-sampling brush to collect cervical cancer cells for screening purposes.
- Standard Letter: Participants received a standard of care letter that tells the participant they are out of date with their cervical cancer screening and should contact their primary care provider to schedule an appointment.
- Total: Total of all reporting groups
Arm/Group | Modified Letter With Self-sampling Request Card | Standard Letter | Total
Number analyzed (Participants) | 333 | 631 | 964
Age, Customized [Number; unit: participants]
  30-65 years | 333 | 631 | 964
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 333 | 631 | 964
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 189 | 359 | 548
  Not Hispanic or Latino | 122 | 239 | 361
  Unknown or Not Reported | 22 | 33 | 55
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 36 | 56 | 92
  White | 82 | 175 | 257
  More than one race | 46 | 80 | 126
  Unknown or Not Reported | 169 | 315 | 484
Region of Enrollment [Number; unit: participants]
  United States | 333 | 631 | 964
Insurance type [Count of Participants; unit: Participants]
  private | 46 | 75 | 121
  other | 267 | 512 | 779
  Missing | 20 | 44 | 64

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Cervical Cancer Screening
Description: To compare the percentage of cervical cancer screenings completed in the control group who received a standard letter with the percentage of cervical cancer screenings completed in the intervention group who receive a modified letter with a self-sampling option.
Time Frame: Three months after the letter is sent.
Measure: Count of Participants; unit: Participants
Groups:
- Modified Letter With Self-sampling Request Card: There were 333 participants in this group. This group received a modified letter telling the participant they are out of date with their cervical cancer screening. They also received information on the self-sampling kit and were provided a card that they can send back to the study team in order to have a kit sent to their house. The kit included a pre-paid mailer so that it can be sent back to the lab for testing. The result were then be shared with the participant.
  Evalyn Self-Sampling Brush: A self-sampling brush to collect cervical cancer cells for screening purposes.
- Standard Letter: There were 631 participants in this group. Participants received a standard of care letter that tells the participant they are out of date with their cervical cancer screening and should contact their primary care provider to schedule an appointment.
Arm/Group | Modified Letter With Self-sampling Request Card | Standard Letter
Number analyzed (Participants) | 333 | 631
Participants | 40 | 95

2. Primary Outcome: Use of the Self-sampling Kit
Description: Evaluate the number of participants request and use the self-sampling kit in the intervention group.
Time Frame: Three months after the letter is sent
Measure: Count of Participants; unit: Participants
Arm/Group | Modified Letter With Self-sampling Request Card
Number analyzed (Participants) | 333
Participants | 2

3. Secondary Outcome: Overall Rate of Cervical Cancer Screening Over Both the Control and Intervention Group
Description: Overall rate of cervical cancer screenings for both the control group and the intervention group.
Time Frame: Three months after the letter is sent
Measure: Count of Participants; unit: Participants
Groups:
- All Participants: Control and Intervention: Combined total participants in both control and intervention arm
Arm/Group | All Participants: Control and Intervention
Number analyzed (Participants) | 964
Participants | 135

ADVERSE EVENTS:
Time Frame: 3 months
Groups:
- Modified Letter With Self-sampling Request Card: This group will receive a modified letter telling the participant they are out of date with their cervical cancer screening. They will also receive information on the self-sampling kit and will be provided a card that they can send back to the study team in order to have a kit sent to their house.
Arm/Group | Modified Letter With Self-sampling Request Card | Standard Letter
All-Cause Mortality (participants affected / at risk) | 0/333 | 0/631
Serious Adverse Events (participants affected / at risk) | 0/333 | 0/631
Other Adverse Events (participants affected / at risk) | 0/333 | 0/631

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-22): https://cdn.clinicaltrials.gov/large-docs/88/NCT04658888/Prot_SAP_000.pdf